CLINICAL TRIAL: NCT05350046
Title: Development of Physical Activity Features for Ear-worn Devices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: 57GGardner (Industry)
Collaborators: Philips BioTelemetry Research (Unknown); Trialfacts (Unknown)
Responsible Party: Sponsor-Investigator, 57GGardner, Principal Investigator, Sonova AG
Organization: Sonova AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRF-485
Record Dates: First submitted 2022-04-21; First posted 2022-04-27 (Actual); Last update posted 2023-12-04 (Actual); Status verified 2023-11

CONDITIONS: Hearing Loss; Well Aging
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Physically active adults (Experimental): A cohort of physically-active adults will use ear-worn prototype devices and established gold standard and comparator devices during rest periods, physical activity, and various activities of daily living.
  Interventions: Device: Ear-worn prototype devices

INTERVENTIONS:
Device: Ear-worn prototype devices — Hearing instrument including sensors to track movement and estimations of biological information.
  Other Names: Phonak Audeo

SUMMARY:
This study incorporates data collection to aid in development of software features related to physical activity for users of ear-worn devices.

DETAILED DESCRIPTION:
This exploratory study involves data collection of adults performing physical activities and activities of daily living for the purpose of comparing data collected by the ear-worn device under test and established gold standard/reference devices and consumer electronic devices. Data collected will be used in the development of software features related to physical activities to benefit the experience of ear-worn device users.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 - 85
* Minimum height 5'3"
* Fully vaccinated against Covid -19
* Willing and able perform various exercise activities at a light and moderate relative intensity, such as riding a stationary bike, walking and jogging on a treadmill, and performing squatting movements.
* Non-smoker for the past 6 months.
* Willing to abstain from caffeine and alcohol 6 hours before participation.
* Willing to fast from eating 4 hours before participation.

Exclusion Criteria:

* History of chronic heart disease or significant cardiac events (e.g. cardiac arrythmia).
* Diagnosed with diabetes mellitus or other metabolic disorder.
* History of cerebral vascular accident.
* History of pulmonary disorder.
* Experiencing orthopedic injury or disorders that restrict movement or cause painful physical activity.
* History of neurodegenerative or neuromuscular pathology.
* Advised by a healthcare professional to not participate in physical activity.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
Accuracy of ear-worn device information | data collection during activities ranging in duration from 5-20 minutes
  Accuracy of information provided by the ear-worn device in comparison to the comparator devices using mean absolute percentage error calculations

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ross, MS, Study Director — Sonova USA Inc
Locations (1):
- Sonova Silicon Valley, Fremont, California, United States

IPD SHARING:
Plan to Share IPD: No